CLINICAL TRIAL: NCT01839630
Title: Study on Transarterial Chemoembolization Combined With Sorafenib in Chinese Patients With Unresectable Hepatocellular Carcinoma (SUCCESS)
Brief Title: Sorafenib Concomitantly Used With TACE (Transarterial Chemoembolization) in uHCC (Unresectable Hepatocellular Carcinoma) Patients in China
Acronym: SUCCESS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16608; NX1216CN (Other: company internal)
Record Dates: First submitted 2012-11-23; First posted 2013-04-25 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Sorafenib; Hepatocellular cancer; TACE combination; Treatment pattern; Safety; Effectiveness
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — sorafenib treatment (including dose, duration, modification) and TACE procedure are decided by the investigator

SUMMARY:
This study is to obtain the characteristics and treatment pattern of the unresectable HCC patients who are candidates for systemic therapy and in whom a decision to treat with sorafenib from early stage of TACE treatment course (concomitantly use no later than the 3rd TACE procedure) has been made under real-life practice conditions.this study will also conclude the safety and effectiveness of combination in uHCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/ cytologically documented or radiographically diagnosed unresectable HCC who are candidates for systemic therapy and for whom a decision to treat with sorafenib has been made. Radiographic diagnosis needs typical findings of HCC by radiographic method i.e. on multi-dimensional dynamic CT, CT hepatic arteriography (CTHA)/CT arterial portography (CTAP) or MRI;
* Patients receive the first dose of sorafenib no later than 1 week (<=7days) after the 3rd TACE procedure
* Patients did not receive other prior systemic treatment by using target therapy
* Patients must sign the informed consent form;
* Patients must have a life expectancy of at least 3 months;
* The physician must be willing to complete and submit all CRFs;
* The physician must be willing to submit to a site audit with verification of source documents and validation of data reported;

Exclusion Criteria:

* The first dose of sorafenib 7 days after the 3nd TACE procedure
* Exclusion criteria must follow the approved local product information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unresectable HCC patients and be candidates for concomitantly systemic therapy with sorafenib + TACE. Considering the local practice and possible clinical benefits, sorafenib should not be initiated later than 7 days after the 3rd TACE course. No prior tartgeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2016-08-06 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Summarized patient characteristics | up to 3 years
  Patient characteristics are hepatic virus infection status, surgery history, tumor size, number of tumor, macroscopic vascular invasion (MVI), extra-hepatic spread (EHS), cirrhosis, ECOG score, Child-Pugh score, BCLC stage, etc.

SECONDARY OUTCOMES:
Number of participants with adverse events( AE) and Serious adverse events(SAE) as a measure of safety and tolorability | up to 3 years
overall survival (OS) by the mRECIST (Modified Response Evaluation Criteria in Solid Tumor) Criteria for treatment of uHCC patients | up to 3 years
progression-free survival (PFS) by the mRECIST for treatment of uHCC patients | up to 3 years
time to progression (TTP) by the mRECIST for treatment of uHCC patients | up to 3 years
response rate (RR) by the mRECIST for treatment of uHCC patients | up to 3 years
Clinical control Rate (DCR) by the mRECIST for treatment of uHCC patients | up to 3 years
Clinical benefit rate (CBR) by the mRECIST for treatment of uHCC patients | up to 3 years
Treatment pattern of Sorafenib | up to 3 years
  Treatment pattern included: Duration and dosage of Sorafenib treatment; reason for Sorafenib dosage modification/discontinuation; anticancer combination therapy; treatment after radiographic relapse; comorbidities and their impact on disease outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, China